CLINICAL TRIAL: NCT02401373
Title: A Phase 1, Dose-escalation, Open Clinical Trial to Evaluate Safety, Tolerability and Immunogenicity of the Recombinant Human Type 5 Adenovirus Vector Based Ebola Vaccine (Ad5-EBOV) in Healthy Adult Africans Aged Between 18-60 Years in China
Brief Title: A Phase I Trial to Evaluate Ad5-EBOV in Healthy Adult Africans in China.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: First Affiliated Hospital of Zhejiang University (Other)
Collaborators: Beijing Institute of Bioengineering, Academy of Military Medical Sciences (Unknown); Tianjin Cansino Biotechnology Inc (Industry)
Responsible Party: Principal Investigator, Lanjuan Li, Academy of Engineering, First Affiliated Hospital of Zhejiang University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: GR2015VCT001
Record Dates: First submitted 2015-03-24; First posted 2015-03-27 (Estimated); Last update posted 2015-07-16 (Estimated); Status verified 2015-07

CONDITIONS: Ebola Virus Disease
Keywords: Vaccines; Ebola Virus Disease
MeSH Terms: conditions — Hemorrhagic Fever, Ebola

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- low dose (Experimental): 30 participants will be firstly recruited and assigned to receive the low dose of Recombinant Human Type 5 Adenovirus Vector Based Ebola Vaccine (Ad5-EBOV).
  Interventions: Biological: Ad5-EBOV
- High dose (Experimental): After the safety of the low dose vaccination is confirmed, another 30 participants will be recruited and assigned to receive the high dose of Recombinant Human Type 5 Adenovirus Vector Based Ebola Vaccine (Ad5-EBOV).
  Interventions: Biological: Ad5-EBOV

INTERVENTIONS:
Biological: Ad5-EBOV — intramuscular injection

SUMMARY:
This is a single center, open, dose-escalation phase 1 clinical trial. This study will determine the safety and side-effect profile, and immunogenicity of an investigational Ad5-EBOV vaccine in Healthy Adult Africans aged between 18-60 years in China.

DETAILED DESCRIPTION:
This is a single center, open, dose-escalation clinical trial. According to the Chinese guidelines for vaccine clinical trial, the sample size of a phase 1 clinical trial should be at least 20. In this study, a total of 60 participants will be included.30 participants will be firstly recruited and assigned to receive the low dose Ad5-EBOV. After the safety of the low dose vaccination is confirmed, another 30 participants will be recruited and assigned to receive the high dose Ad5-EBOV.

The whole follow-up period for each participant will be 28 days.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 18 and 60 years.
* African in China.
* Able to understand the content of informed consent and willing to sign the informed consent
* Able and willing to complete all the secluded study process during the whole study follow-up period (about 1 month).
* A body mass index (BMI) 18.5-35.0 kg/m2
* Hemoglobin ≥110g/L for female, and ≥120g/L for male.
* White blood cells (WBC) 4.0-10.0×109 cells/L
* Total lymphocyte Count 0.8-4.5×109 cells/L
* Platelets 100-300×109 cells/L
* Alanine aminotransferase (ALT) 0-40U/L
* Serum creatinine 44-106μmol/L
* Active partial thromboplastin time (APTT) 20-40 seconds
* Prothrombin time (PT) 10-14 seconds
* Negative in HIV diagnostic blood test
* Axillary temperature ≤37.0°C on the day of enrollment
* General good health as established by medical history and physical examination.

Exclusion Criteria:

* Family history of seizure, epilepsy, brain or mental disease
* Participant that has a medical history of any of the following: allergic history of any vaccination or drugs, or allergic to any ingredient of the Ad5-EBOV, such as mannitol.
* Woman who is pregnant, breast-feeding or positive in β-HCG (human chorionic gonadotropin) pregnancy test (urine) on day of enrollment, or become pregnant during the next 6 months
* Any acute fever disease or infections in last 7 days
* Major congenital defects or not well-controlled chronic illness, such as asthma, diabetes, or thyroid disease
* Hereditary angioneurotic edema or acquired angioneurotic edema
* Urticaria in last one year
* Asplenia or functional asplenia
* Platelet disorder or other bleeding disorder may cause injection contraindication
* Faint at the sight of blood or needles.
* Prior administration of immunodepressant or corticosteroids, antianaphylaxis treatment, cytotoxic treatment in last 6 months
* Prior administration of blood products in last 4 months
* Prior administration of other research medicines in last 1 month
* Prior administration of attenuated vaccine in last 1 month
* Prior administration of inactivated vaccine in last 14 days
* Current anti-tuberculosis prophylaxis or therapy
* Any condition that in the opinion of the investigators may interfere with the evaluation of study objectives

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 61 (Actual)
Dates: Start 2015-03; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
A Phase I, Open Clinical Trial to Evaluate the Adenovirus Type 5 Vector Based Ebola Virus Disease Vaccine (Ad5-EBOV) in Healthy Adult Africans in China. | From March to July, 2015

CONTACTS AND LOCATIONS:
Overall Officials: Lanjuan Li, Principal Investigator — First Affiliated Hospital of Zhejiang University
Locations (1):
- First affiliated hospital of Zhejiang University, Hangzhou, Zhejiang, China

REFERENCES:
- [Derived] Wu L, Zhang Z, Gao H, Li Y, Hou L, Yao H, Wu S, Liu J, Wang L, Zhai Y, Ou H, Lin M, Wu X, Liu J, Lang G, Xin Q, Wu G, Luo L, Liu P, Shentu J, Wu N, Sheng J, Qiu Y, Chen W, Li L. Open-label phase I clinical trial of Ad5-EBOV in Africans in China. Hum Vaccin Immunother. 2017 Sep 2;13(9):2078-2085. doi: 10.1080/21645515.2017.1342021. Epub 2017 Jul 14. PMID 28708962